CLINICAL TRIAL: NCT01534910
Title: Effect of Aged Garlic Extract on Atherosclerosis
Acronym: Garlic4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21567-01
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Metabolic Syndrome
Keywords: garlic; ct angiography; atherosclerosis; carotid IMT
MeSH Terms: conditions — Metabolic Syndrome; Atherosclerosis | interventions — kyolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator): placebo
  Interventions: Drug: placebo
- Aged Garlic Extract (Active Comparator): 2400 mg of aged garlic extract
  Interventions: Drug: aged garlic extract

INTERVENTIONS:
Drug: aged garlic extract — 2400 mg a day
  Other Names: Kyolic
  Arms: Aged Garlic Extract
Drug: placebo — placebo
  Arms: Sugar pill

SUMMARY:
The investigators will be assessing the effect of Aged Garlic Extract on the coronary arteries. The investigators will enroll patients in a double blind study, where half the patients will receive placebo, and have the patients undergo a series of tests of plaque (CT scan of the heart, carotid ultrasound) and follow the patients on the drug or placebo and then repeat the tests and blood work at the end of one year. The investigators will assess if being on aged garlic extract adds any benefit to plaque in the coronary or neck arteries. The investigators will also assess the effect of aged garlic extract on markers of inflammation. Patients will receive free drug, free testing and be compensated, and learn more about their heart and neck arteries. if successful, more patients can use this drug to benefit their health. The harms include the radiation from the CT scan and the medication, which has mild side effects.

DETAILED DESCRIPTION:
The investigators will be assessing the effect of Aged Garlic Extract on the coronary arteries. The investigators will enroll patients in a double blind study, where half the patients will receive placebo, and have the patients undergo a series of tests of plaque (CT scan of the heart, carotid ultrasound) and follow the patients on the drug or placebo and then repeat the tests and blood work at the end of one year. The investigators will assess if being on aged garlic extract adds any benefit to plaque in the coronary or neck arteries. The investigators will also assess the effect of aged garlic extract on markers of inflammation. Patients will receive free drug, free testing and be compensated, and learn more about their heart and neck arteries. if successful, more patients can use this drug to benefit their health. The harms include the radiation from the CT scan and the medication, which has mild side effects. The study will perform advanced CT angiography at baseline and follow up along with carotid intimal media thickness testing, to see if plaque is slowed down by Aged Garlic Extract

ELIGIBILITY:
Inclusion Criteria

* Age 40-65 years
* Framingham risk score 6-20%, and at least 2 components of the metabolic syndrome as defined by ATP III Clinical Identification of the Metabolic Syndrome (including impaired fasting glucose > 110 mg/dl, treated hypertension or SBP > 130 or DBP > 85 mm Hg, plasma triglycerides > 150 mg/dl, HDL cholesterol < 35 mg/dl for men or < 40 mg/dl for women, abdominal obesity as defined as waist > 40 in for men, > 35 in for women)
* Subjects must provide written informed consent after the scope and nature of the investigation has been explained to them
* Subjects should be stable on their concomitant medications for at least 26 weeks prior to randomization
* Calcium Score > 20 at baseline
* Subjects who agree to refrain from other anti-glycemic agent Exclusion Criteria
* A contraindication to AGE including: known hypersensitivity to drug.
* Any unstable medical, psychiatric or substance abuse disorder that in the opinion of the investigator or principal investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
* Weight in excess of 300 pounds
* Bleeding disorder
* History of known coronary artery disease, myocardial infarction, stroke or life-threatening arrhythmia within the prior six months
* NYHA Class II- IV heart failure
* History of malignancy within the last 5 years (other than skin cancer) or evidence of active cancer which would require concomitant cancer chemotherapy
* Serum creatinine > 1.4 mg/dl
* Diabetes Mellitus
* Triglycerides > 400 at visit 1
* Drug or alcohol abuse, or current intake of more than 14 standard drinks per week
* Concurrent enrollment in another placebo-controlled trial
* Partial ileal bypass or known gastrointestinal disease limiting drug absorption
* Current diabetes or intake of anti-diabetic or other prohibited drug
* Current tobacco use
* Current use of anticoagulants (except for anti-platelet agents)
* Renal failure
* History of hypertensive encephalopathy or cerebrovascular accident
* Hematological or biochemical values at screening outside the reference ranges considered as clinically significant in the opinion of the investigator or PI

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Budoff, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matsumoto S, Nakanishi R, Li D, Alani A, Rezaeian P, Prabhu S, Abraham J, Fahmy MA, Dailing C, Flores F, Hamal S, Broersen A, Kitslaar PH, Budoff MJ. Aged Garlic Extract Reduces Low Attenuation Plaque in Coronary Arteries of Patients with Metabolic Syndrome in a Prospective Randomized Double-Blind Study. J Nutr. 2016 Feb;146(2):427S-432S. doi: 10.3945/jn.114.202424. Epub 2016 Jan 13. PMID 26764322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all 65 participants were recruited
Period: Overall Study
Arm/Group | Sugar Pill | Aged Garlic Extract
Started | 33 | 32
Completed | 29 | 28
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Sugar Pill: placebo
  placebo: placebo patients were randomized to placebo
- Aged Garlic Extract: 2400 mg of aged garlic extract
  aged garlic extract: 2400 mg a day patients randomized to aged garlic extract
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Aged Garlic Extract | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (7) | 56 (8) | 57 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: CT Angiography Plaque
Description: we will measure low attenuation plaque at baseline (in volume) and then again at 1 year. we will assess if there is a reduction in low attenuation plaque volume (percent change from baseline), defined as [followup-baseline]/baseline x100%.
  Baseline was time zero, followup CT scan was 1 year.
Time Frame: baseline to 1 year
Measure: Mean (Standard Deviation); unit: percent change of low attenuation plaque
Groups:
- Sugar Pill: placebo
  placebo: placebo patients were randomized to placebo No adverse events
- Aged Garlic Extract: 2400 mg of aged garlic extract
  aged garlic extract: 2400 mg a day patients randomized to aged garlic extract No adverse events
Arm/Group | Sugar Pill | Aged Garlic Extract
Number analyzed (Participants) | 28 | 27
percent change of low attenuation plaque | 0.17 (1.97) | -1.53 (2.32)

2. Secondary Outcome: Coronary Calcium
Description: Agatston score is a semi-automated tool to calculate a score based on the extent of coronary artery calcification detected by an unenhanced low-dose CT scan. The calculation is based on the weighted density score given to the highest attenuation value (HU) multiplied by area of the calcification speck. The grading of coronary artery disease (based on total calcium score) is as follows: no evidence of CAD: 0 calcium score, minimal: 1-10, mild: 11-100, moderate: 101-400, and severe: >400
Time Frame: 1 year
Population: patients undergoing two calcium scores
Measure: Mean (95% Confidence Interval); unit: agatston units
Arm/Group | Sugar Pill | Aged Garlic Extract
Number analyzed (Participants) | 28 | 27
agatston units | 95 [74 to 116] | 49 [20 to 78]

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Aged Garlic Extract
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No